CLINICAL TRIAL: NCT03493893
Title: 10 Year Review of the Experience of the PFNA ,TFNA the Affixus Nail
Status: Completed | Type: Observational
Sponsor: Princess Alexandra Hospital, Brisbane, Australia (Other)
Responsible Party: Principal Investigator, Genni Lynch, Research coordinator, Princess Alexandra Hospital, Brisbane, Australia
Other Study IDs: 123456
Record Dates: First submitted 2017-04-10; First posted 2018-04-11 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Fractured Neck of Femur
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Affixus: To compare Affixus to PFNA and TFNA
  Interventions: Device: Intermedullary nail
- PFNA: To compare PFNA to Affixus and TFNA
  Interventions: Device: Intermedullary nail
- TFNA: To compare TFNA toPFNA and Affixus
  Interventions: Device: Intermedullary nail

INTERVENTIONS:
Device: Intermedullary nail — investigate the clinical effects of these design changes from the use of three different IM nail designs in the management of extracapsular hip fractures.
  Other Names: Affixus, PFNA, TFNA

SUMMARY:
The aim of this study was to investigate the clinical effects of design changes from the use of three different IM nail designs in the management of extracapsular hip fractures.

DETAILED DESCRIPTION:
Intertrochanteric hip fractures are one of the more common orthopaedic presentations, with an approximate incidence in Australia of 230 cases per 100,000 population. The importance of this pathology is well documented being the major fracture-related health care cost and cause of mortality in all sexes over 50 years of age.

Contemporary fixation of the proximal femur is performed utilising a number of implants adopting different concepts and techniques. Cephalomedullary/Intermedullary femoral nails (IM nails) over the last 15 years have gained popularity. IM nails are implanted via a small incision and intermedullary insertion through the greater trochanter, secured by passing a screw or blade through the femoral neck into the femoral head. This nailing technique offers the theoretical benefits of a smaller incision with less tissue dissection and hence reduced blood loss, infection and operating time. As well as a proposed biomechanical advantage due to a shorter lever arm, sharing the load and minimising proximal collapse.

Biomechanical studies of IM nails in the use of extracapsular fractures of the femoral neck have found benefit over existing sliding/compression hip screws (CHS). Advantages have been observed in combined bending and compression performance to failure. As well as postoperative rigidity in unstable subtrochanteric fractures, and load bearing capability. Significantly greater fatigue strength and fatigue life have additionally been shown in cyclic loading assessment and reduced incidence of cut out has been observed, showing benefit over the use of CHS.

Early trials however found a higher rate of operative complications involving IM fixation, including fractures at the tip of the nail or related to distal locking. Following this several studies have compared the clinical outcomes of CHS vs IM nails with varying findings questioning the overall patient benefit, especially in stable fracture patterns. From a review of the past literature the common trend is a longer operative time and higher associated blood loss with CHS, but fewer intraoperative surgical related complications and less fluoroscopic time with the use of nails. IM nail use has shown to offer better post-operative ambulatory function and reduced limb shortening but it appears due to the early complications of this technique numerous variations in implant design have emerged.

Purpose In recent years further development has occurred in nail design in an attempt to reduce the incidence of fixation failure. The aim of this study was to investigate the clinical effects of these design changes from the use of three different IM nail designs in the management of extracapsular hip fractures.

ELIGIBILITY:
Inclusion Criteria:

. fractured neck of femur

Exclusion Criteria:

. NOT fractured neck of femur

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Reoperation | 12 months
  Taken back to the operating room for reoperation

SECONDARY OUTCOMES:
Failure | 12 months
  Unable to weight bear

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Cooke, Principal Investigator — Princess Alexandra Hospital

IPD SHARING:
Plan to Share IPD: No